CLINICAL TRIAL: NCT01959919
Title: Non Interventional Longitudinal Study To Assess The Acceptability And The Satisfaction Of Patients With Haemophilia A Treated Both On Demand And On Prophylaxis With A New Factor Viii Delivery System Fusengo
Brief Title: Evaluation Of Acceptability And Satisfaction Of Hemophilia Patients Treated With FusENGO
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1831081
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1: Device
  Interventions: Device: Refacto FusENGO

INTERVENTIONS:
Device: Refacto FusENGO — Dosage will be chosen by PI based on patient condition.

SUMMARY:
This study aims to investigate prospectively throughout a period of 3- 6 months and not to exceed 12 months (according to local therapeutic plans) patients experiences of treatment with Factor VIII in the new device named FuseNGO, a new delivery system for Factor VIII compared to their previous delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Male adults (aged 18 to 65 years) with Haemophilia A (all severity levels) who currently use FVIII treatment either prophylactically or on-demand using traditional factor VIII delivery mechanisms.
* Patients advised for any reason by their physician to switch to a new factor VIII delivery device, namely FuseNGO, before receiving any details about this study or Patients who requested to be treated with a new factor VIII delivery device namely FuseNGO, before receiving any details about this study.

Exclusion Criteria:

* Patients not previously recommended by their physician to switch to this new factor VIII delivery system or Patients who did not previously ask their physician to be switched to this new factor VIII delivery system.
* Patients for which it is anticipated that 10 infusions will not occur in the 12 months following their inclusion in the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Approximately 200 patients with Hemophilia A (all severity levels) will be enrolled in approximately 20 centers in Italy.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- Italy (19):
  - Istituto di Ematologia, Rome, Lazio
  - Ospedale SS. Annunziata - USL 1, Sassari, Sardinia
  - Azienda Ospedale Policlinico Consorziale, Bari
  - Struttura Complessa Di Oncoematologia Pediatrica E Patologia Della Coagulzione, Cagliari
  - Ospedale Ferrarrotto, Catania
  - Azienda Ospedaliera Ciaccio - Ospedale Pugliese, Catanzaro
  - Azienda Ospedaliera Careggi, Florence
  - Centro regionale di diagnosi e trattamento dell'Emofilia e delle malattie dell'emostasi e trombosi, Macerata
  - Ospedale Maggiore Policlinico Mangiagalli E Regina Elena, Milan
  - Dipartimento Medicina Clinica e Sperimentale, Napoli
  - Centro Emofilia e Trombosi - Centro delle Microcitemie, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Policlinico P Giaccone, Palermo
  - Arcispedale S. Maria Nuova, AO di Reggio Emilia, Reggio Emilia
  - Policlinico Agostino Gemelli, Rome
  - Ospedale Molinette, Torino
  - SC Servizio Immunotrasfusionale, Torino
  - SOS Malattie Emorragiche e Trombotiche AOU "S.M.M." Udine, Udine
  - Anna Chiara Giuffrida, Verona

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1831081&StudyName=Evaluation%20Of%20Acceptability%20And%20Satisfaction%20Of%20Hemophilia%20Patients%20Treated%20With%20FusENGO

RESULTS

PARTICIPANT FLOW:
Groups:
- Refacto AF FuseNGo: Participants with haemophilia A, who were receiving clotting factor VIII treatment prior to enrollment in this study, used Refacto AF FuseNGo (intravenous infusion of moroctocog alfa, a human recombinant clotting factor VIII, delivered by system FuseNGo) either prophylactically or on-demand and were observed for maximum up to Week 52. Dosage and use of Refacto AF FuseNGo was based on investigator's judgement according to approved summary of product characteristics (SmPC).
Period: Overall Study
Arm/Group | Refacto AF FuseNGo
Started | 86
Completed | 84
Not Completed | 2
Not completed — Did not meet the eligibility criteria | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all the participants who were enrolled and received at least 1 dose of Refacto AF FuseNGo.
Groups:
- Refacto AF FuseNGo: Participants with haemophilia A, who were receiving clotting factor VIII treatment prior to enrollment in this study, used Refacto AF FuseNGo (intravenous infusion of moroctocog alfa, a human recombinant clotting factor VIII, delivered by system FuseNGo) either prophylactically or on-demand and were observed for maximum up to Week 52. Dosage and use of Refacto AF FuseNGo was based on investigator's judgement according to approved SmPC.
Arm/Group | Refacto AF FuseNGo
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.99 (11.206)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 86
Time for Reconstructing the Drug [Mean (Standard Deviation); unit: minutes] — In this parameter time consumed for performing steps to reconstitute the drug prior to infusion of drug is reported.
  minutes | 10.79 (7.419)
Burden of Clotting Factor Treatment Score [Mean (Standard Deviation); unit: units on scale] — HaemoPREF is a participant rated 14-item instrument to measure experience of clotting factor treatment for determining the score for burden of clotting factor treatment, 2 items were assessed by participants: 1) time consumption to treat with treatment and 2) difficulty in finding vein to inject treatment in to. Each of the 2 items was scored on a scale of 0 (most difficult) to 20 (least difficult) and summed up to give a total overall score range of 0 (most burdened) to 40 (least burdened). Higher scores indicate a lower burden of treatment.
  units on scale | 11.88 (4.652)
Impact of Clotting Factor Treatment Score [Mean (Standard Deviation); unit: units on scale] — HaemoPREF is a 14-item instrument to measure experience of clotting factor treatment. For score for impact of clotting factor treatment, 3 items were assessed by participants: 1)difficulty to travel for holidays or works, 2)difficulty to perform daily activities including work or study and 3)difficulty to perform social or leisure activities. Each of 3 items was scored on a scale of 0(most challenging) to 10(least challenging), and summed up to give total overall score range of 0(greatest negative impact) to 30(least negative impact). Higher scores indicate less negative impact on daily life.
  units on scale | 17.86 (7.117)
Risk Associated With Clotting Factor Treatment Score [Mean (Standard Deviation); unit: units on scale] — HaemoPREF is 14-item instrument to measure experience of clotting factor treatment. For score for risk associated with clotting factor treatment,3 items were assessed by participants: 1)worried about getting infected with other disease while on treatment,2)worried to infect treatment while preparing for injection and 3)worried to inject treatment by own. Each of 3 items was scored on a scale of 0(most concerned) to 10(not at all concerned),summed up to give total overall score range of 0(most worried) to 30(least worried). Higher scores indicate lower levels of worry associated with treatment.
  units on scale | 19.69 (7.076)

OUTCOME MEASURES:

1. Primary Outcome: Ease of Using Clotting Factor Treatment Score
Description: HaemoPREF is a participant rated 14-item instrument to measure experience of clotting factor treatment including ease of use, burden, impact, risk and influence of others on treatment choices. For determining score for ease of using clotting factor treatment, 4 items assessed by participants were: 1) ease to prepare treatment for injection, 2) ease to store treatment, 3) ease to dispose of containers, syringe and needle once used and 4) ease to use current treatment. Each of the 4 items was scored on a scale of 0 (not at all easy) to 10 (extremely easy), and were summed up, to give a total overall score range of 0 (no ease) to 40 (maximum ease). Higher scores indicate greater ease in using clotting factor treatment.
Time Frame: Final Visit (Month 8)
Population: Per-protocol population included all participants who received at least 1 treatment using the Refacto AF FuseNGo and completed the two final questionnaires.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refacto AF FuseNGo
Number analyzed (Participants) | 84
units on a scale | 31.15 (6.539)
Statistical Analysis 1: Comparison: Refacto AF FuseNGo; Comparison between ease of using clotting factor treatment score at Final visit (Month 8) and baseline visit; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test; Mean Difference (Final Values) = -4.907

2. Primary Outcome: Time for Reconstructing the Drug
Description: In this outcome measure time consumed for performing steps to reconstitute the drug prior to infusion of drug is reported.
Time Frame: Final Visit (Month 8)
Population: Per-protocol population all participants who received at least 1 treatment using the Refacto AF FuseNGo and completed the two final questionnaires. Here "Number of Participants Analyzed (N)" signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Refacto AF FuseNGo
Number analyzed (Participants) | 83
minutes | 6.247 (4.3409)
Statistical Analysis 1: Comparison: Refacto AF FuseNGo; Comparison between time for reconstructing the drug at Final visit (Month 8) and baseline visit; Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Final Values) = 4.572, 95% CI 2-sided [3.411 to 5.733], Standard Error of Mean 0.584

3. Primary Outcome: Burden of Clotting Factor Treatment Score
Description: HaemoPREF is a participant rated 14-item instrument to measure experience of clotting factor treatment including ease of use, burden, impact, risk and influence of others on treatment choices. For determining the score for burden of clotting factor treatment, 2 items were assessed by participants: 1) time consumption to treat with treatment and 2) difficulty in finding vein to inject treatment in to. Each of the 2 items was scored on a scale of 0 (most difficult) to 20 ( least difficult) and summed up to give a total overall score range of 0 (most burdened) to 40 (least burdened). Higher scores indicate a lower burden of treatment.
Time Frame: Final Visit (Month 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Refacto AF FuseNGo
Number analyzed (Participants) | 84
units on scale | 13.55 (4.275)
Statistical Analysis 1: Comparison: Refacto AF FuseNGo; Comparison between burden of clotting factor treatment score at Final Visit Month 8 and baseline visit; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test; Median Difference (Final Values) = -3.789

4. Primary Outcome: Impact of Clotting Factor Treatment Score
Description: HaemoPREF is a participant rated 14-item instrument to measure experience of clotting factor treatment including ease of use, burden, impact, risk and influence of others on treatment choices. For determining score for impact of clotting factor treatment, 3 items were assessed by participants: 1) difficulty to travel for holidays or works, 2) difficulty to perform daily activities including work or study and 3) difficulty to perform social or leisure activities. Each of the 3 items was scored on a scale of 0 (most challenging) to 10 (least challenging), and summed up to give a total overall score range of 0 (greatest negative impact) to 30 (least negative impact). Higher scores indicate less negative impact on daily life.
Time Frame: Final Visit (Month 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Refacto AF FuseNGo
Number analyzed (Participants) | 84
units on scale | 20.15 (6.167)
Statistical Analysis 1: Comparison: Refacto AF FuseNGo; Comparison between impact of clotting factor treatment score at Final Visit Month 8 and baseline visit; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test; Median Difference (Final Values) = -3.980

5. Primary Outcome: Risk Associated With Clotting Factor Treatment Score
Description: HaemoPREF is a participant rated 14-item instrument to measure experience of clotting factor treatment including ease of use, burden, impact, risk and influence of others on treatment choices. For determining score for risk associated with clotting factor treatment, 3 items were assessed by participants: 1) worried about getting infected with other disease while using the treatment, 2) worried to contaminate the treatment while preparing for injection and 3) worried to inject treatment by own. Each of the 3 items was scored on a scale of 0 (most concerned) to 10 (not at all concerned), and summed up to give a total overall score range of 0 (most worried) to 30 (least worried). Higher scores indicate lower levels of worry associated with treatment.
Time Frame: Final Visit (Month 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Refacto AF FuseNGo
Number analyzed (Participants) | 84
units on scale | 21.40 (6.733)
Statistical Analysis 1: Comparison: Refacto AF FuseNGo; Comparison between risk associated with clotting factor treatment score at Final Visit Month 8 and baseline visit; Test type: Superiority or Other; p = 0.001, Wilcoxon Signed Ranks Test; Median Difference (Final Values) = -3.445

6. Primary Outcome: Overall Satisfaction Score With Refacto AF FuseNGO
Description: HaemoPREF: participant rated 14-item instrument to measure experience of clotting factor treatment. 14 items: 1) ease to prepare treatment for injection, 2) ease to store treatment, 3) ease to dispose container, syringe, needle once used and 4) ease to use treatment, 5) time consumed with treatment, 6) difficulty in finding a vein to inject treatment, 7) difficulty to travel, 8) difficulty to do daily activities, 9) difficulty to do social or leisure activities, 10) worried for getting infected with other disease while using the treatment, 11) worried to contaminate the treatment while preparing for injection, 12) worried to inject by own, 13) importance of family's opinion to use treatment, 14) importance what others use for their hemophilia. Each item was scaled from 0 (no satisfaction) to 10 (maximum satisfaction). Overall satisfaction score was the sum of 14 items, ranged from 0 (no satisfaction) to 140 (maximum satisfaction). Higher scores indicate greater treatment satisfaction.
Time Frame: Final Visit (Month 8)
Population: Per-protocol population included all participants who received at least 1 treatment using the Refacto AF FuseNGo and completed the two final questionnaires. Here "N" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refacto AF FuseNGo
Number analyzed (Participants) | 83
units on a scale | 93.90 (18.883)

7. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received treatment using Refacto AF Fusnego without regard to possibility of causal relationship. Serious adverse event was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to 28 days after last dose of drug (up to Month 12)
Population: Safety population included all the participants who were enrolled and received at least 1 dose of Refacto AF FuseNGO.
Measure: Number; unit: participants
Arm/Group | Refacto AF FuseNGo
Number analyzed (Participants) | 86
participants
  Adverse Events | 3
  Serious Adverse Events | 0

ADVERSE EVENTS:
Description: Safety population included all the participants who were enrolled and received at least 1 dose of Refacto AF FuseNGo.
Arm/Group | Refacto AF FuseNGo
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 3/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Refacto AF FuseNGo (N=86)
Gastroentheritis (Infections and infestations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
High fever (Bronchitis) (Infections and infestations) | 1
Esophageal varices (Gastrointestinal disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Insomnia and nightmares (Psychiatric disorders) | 1
Flu (Infections and infestations) | 1
Pulpitis (Infections and infestations) | 1
Anal bleeding from hemorrhoids (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
The outcome measure 'ease of storing clotting factor treatment score' was not analyzed as per change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/ termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.